CLINICAL TRIAL: NCT01460498
Title: Phase I-II Study of Low-Dose Azacitidine (Vidaza) in Patients With Chronic Myeloid Leukemia Who Have Minimal Residual Disease While Receiving Therapy With Tyrosine Kinase Inhibitors (VZ-CML-PI-0236)
Brief Title: Azacitidine (AZA) in Minimal Residual Disease (MRD) Chronic Myeloid Leukemia (CML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0254; NCI-2011-03531 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Myeloid Leukemia; CML; Complete cytogenetic remission; CCyR; Minimal residual disease; Philadelphia chromosome (Ph)-; BCR/ABL-positive; Tyrosine kinase inhibitor; TKI; Azacitidine; 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasm, Residual; Philadelphia Chromosome | interventions — Azacitidine; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Group (AZA) (Experimental): Azacitidine (AZA) starting dose 50 mg/m2 a day for 3 days subcutaneous or intravenous of 28 day cycle. TKI at dose received during last 6 months.
  Interventions: Drug: Azacitidine (AZA); Drug: Tyrosine kinase inhibitor (TKI)
- Expansion Group (AZA MTD) (Experimental): Dose Escalation Group plus additional 36 participants for Azacitidine 75 mg/m2 (or Phase I MTD) either subcutaneous or intravenous every day for 3 days of 28 day cycle. TKI at dose received during last 6 months.
  Interventions: Drug: Tyrosine kinase inhibitor (TKI); Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine (AZA) — Starting Dose 50 mg/m2 by subcutaneous or by vein for 3 days of a 28 day cycle.
  Other Names: 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Dose Escalation Group (AZA)
Drug: Tyrosine kinase inhibitor (TKI) — Continuation of dose already receiving during previous 6 months.
Drug: Azacitidine — 75 mg/m2 daily for 3 days, unless MTD defined at lower dose level in Phase I then that would become dose used for Phase II.
  Other Names: 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Expansion Group (AZA MTD)

SUMMARY:
This is a 2 part study. The goal of the first part of this clinical research study is to find the highest tolerable dose of azacitidine that can be given with a TKI that you are already taking (such as Gleevec, Sprycel, or Tasigna). The safety of this drug will also be studied. The goal of the second part is to see if this combination may improve your response to the TKI you are already taking.

Azacitidine is designed to change genes that are thought to cause leukemia. By changing these genes, the drug may help to stop them from causing the disease to grow.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will continue receiving the same TKI at the dose you had been receiving for the last 6 months.

You will receive azacitidine either as an injection under your skin or through a vein every day for 3 to 7 days of each 28-day cycle. The dose and how often you take the drug will depend on when you enter the study. The study staff will tell you how often you will receive the drug.

In the first part of the study, you will be assigned to a dose level of azacitidine based on when you join this study. Up to 2 dose levels of azacitidine will be tested. At least 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. The next group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of azacitidine is found. This is called the Dose Escalation Group.

Once the highest tolerated dose has been found, an extra 36 participants will receive azacitidine at this dose level. This is called the Expansion Group.

If you have severe side effects from the study drug, the study doctor may decide to reduce and/or stop drug dosing until your side effects improve. If the doctor thinks it is in you best interest, your dose may be increased.

Study Visits:

At every visit, you will be asked about any side effects you have had and to list any drugs you may be taking.

* Every 1-2 weeks for 8 weeks, then at the start of every cycle, blood (about 1 teaspoon) will be drawn for routine tests.
* Every 2-4 weeks for 8 weeks, then before each cycle, blood (about 1 teaspoon) will also be drawn to test your kidney and liver function.
* Before each cycle for 3 cycles, then every 3-6 cycles until 1 year, then every 6-12 cycles, blood (about 1 tablespoon) drawn for molecular testing.
* Every 3-6 months in Year 1, then as often the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease.
* If you are in the Expansion Group, every 3 months (+/- 1 month) for the first 6 months, then every 6-12 months, you will have a complete physical exam.
* If you are in the Dose Escalation Group, every 2 weeks for the first month, Months 1, 2, 3, and 6 (+/- 1 month), and then every 6-12 months, you will have a complete physical exam.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment and follow-up visits.

This is an investigational study. TKIs are approved for the treatment of CML. Azacitidine is FDA approved and commercially available for the treatment of patients with MDS. The combination of these drugs to treat CML is investigational.

Up to 48 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 16 years or older with Philadelphia chromosome (Ph)- or BCR/ABL-positive CML (as determined by cytogenetics, FISH, or PCR).
2. Patients must have received FDA-approved TKI therapy for at least 18 months and not have increased their dose of FDA-approved TKI in the last 6 months. Patients participating on frontline protocols 2005-0048 (nilotinib) and 2005-0422 (dasatinib) are eligible for enrollment on this study.
3. Phase II patients must be in complete cytogenetic remission. For the phase I portion of the study, patients may be included without a complete cytogenetic remission provided they are in chronic phase.
4. Phase II patients must have detectable BCR-ABL transcript levels meeting at least one of the following criteria: Patient has never achieved a major molecular response, and transcript levels have shown in at least two consecutive measures separated by at least 1 month to have increased by any value, or Achieved a major molecular response that has been lost with an increase in transcript levels by at least 1-log, confirmed in two consecutive analyses separated by at least 1 month, or The patient has received therapy for at least 2 years and does not have a sustained major molecular response, or The patient has received therapy for at least 5 years and does not have a sustained complete molecular response. Patients included in the phase I portion of the study are eligible regardless of their level of BCR-ABL transcripts.
5. Patients must not have had a known continuous interruption of imatinib therapy of greater than 14 days or for a total of 6 weeks in the 6 months prior to enrollment.
6. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.
7. ECOG performance status </= 2.
8. Adequate organ function defined as: bilirubin < 2x upper limit of normal (ULN) (unless associated with Gilbert's syndrome), and ALT or AST </= 2.5x ULN.
9. ANC >/=1 x10(9)/L and platelets >/= 50 x10(9)/L.
10. Serum creatinine < 1.8 mg/dL or creatinine clearance greater or equal than 40 cc/min as defined by the Cockcroft-Gault Equation*. Males(mL/min):(140-age)* ABW(kg) / 72* (serum creatinine(mg/dl)); Females (mL/min):0.85*(140-age)* ABW(kg) / 72*(serum creatinine (mg/dl))
11. Women of childbearing potential should be advised to avoid becoming pregnant and practice effective methods of contraception. Men should be advised not to father a child while receiving treatment with azacitidine. Azacitidine is classified as Pregnancy Category D. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study.
12. Women of childbearing potential should have a pregnancy test within 7 days before initiation of study drug.

Exclusion Criteria:

1. Patients receiving any other investigational agents.
2. Patients who are pregnant or breast-feeding.
3. Patients with clinically significant heart disease (NYHA Class III or IV).
4. Known or suspected hypersensitivity to azacitidine or mannitol.
5. Patients with advanced malignant hepatic tumors.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Azacitidine | First 28 day cycle
  MTD is defined as the highest dose level in which 6 patients have been treated and one or fewer patient experiences Dose-Limiting Toxicity (DLT) within the first course of treatment.
Number of Participants with Decrease of Transcript Levels by at Least One Log (or Undetectable Transcript Level) Within 12 Months | Baseline to 12 months
  Participants with response defined as a greater than a one-log reduction of BCR-ABL transcript levels from the baseline level at the time vaccination was initiated, or a disappearance of BCR-ABL transcripts (i.e., complete molecular response) within 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT01460498/Prot_SAP_000.pdf